CLINICAL TRIAL: NCT03395574
Title: Effect of Terlipressin on Cerebral Oxygen Saturation and Cerebral Blood Flow During Living Donor Liver Transplantation
Brief Title: Effect of Terlipressin on Cerebral Oxygen Saturation During Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-113-2017
Record Dates: First submitted 2017-12-25; First posted 2018-01-10 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Terlipressin Adverse Reaction; Liver Transplantation
MeSH Terms: interventions — Terlipressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- terlipressin group (Experimental): group will receive terlipressin infusion one mg in 50 ml normal saline will be given over 30 minute as loading dose then will be maintained as infusion of 160 μg per hour (8 ml/h).
  Interventions: Drug: Terlipressin
- saline (control) group (Placebo Comparator): group will receive normal saline infusion 50 ml normal saline will be given over 30 minute as loading dose then will be maintained as infusion of (8 ml/h).
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Terlipressin — drug will be given after 30 minutes of induction of anesthesia
  Arms: terlipressin group
Drug: Normal saline — drug will be given after 30 minutes as placebo in control group
  Arms: saline (control) group

SUMMARY:
in our study the investigators aim to assess the effect of terlipressin on cerebral oxygenation monitored by cerebral oxymetry and cerebral blood flow measured by transcranial doppler.

DETAILED DESCRIPTION:
All patients will receive 6ml /kg/h Ringer acetate solution as a maintenance intraoperative fluid. If pulse pressure variations (PPV) is more than 15%, the patient will be considered as fluid responder and will receive a 250-ml bolus of albumin 5% to maintain PPV ≤15%. Blood transfusion will be given based on a hemoglobin level (< 7 g/dl) in both (control group) and (terlipressin group). Other blood products will be transfused guided by lab result; Fresh frozen plasma will be given when INR > 2 and platelets will be given when platelets <30.000/mm3. The patients will be randomly allocated into 2 groups; Group T (Terlipressin group) and group S (Normal saline 0.9%).

For (terlipressin group) all patients will receive loading dose of terlipressin (1mg diluted with 50 ml of normal saline 0.9% solution over 30 min) and it will be maintained by continuous infusion at rate of 160 μg per hour (8 ml/h).

For (control group) all patient will receive 50 ml of normal saline 0.9% solution over 30 min and will be maintained continuous infusion at rate of 8 ml/h.

Drugs will be prepared by the nurse and the investigator will be blinded to the drug given.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-IV undergoing orthotopic liver transplantation.
* Age above 18 years.

Exclusion Criteria:

* Age below 18 years.
* Patients on Terlipressin preoperative.
* Patients known allergic to Terlipressin.
* Portal vein thrombosis.
* Ischemic heart disease.
* Patients with T. bilirubin level above 7 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
cerebral oxygen saturation | one hour after infusion of drug
  regional oxygen saturation assessed by cerebral oxymetry with probes applied on forehead

SECONDARY OUTCOMES:
cerebral oxygen saturation | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  regional oxygen saturation assessed by cerebral oxymetry with probes applied on forehead
resistive index of middle cerebral artery | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by trans cranial Doppler
peak velocity, end diastolic velocity of middle cerebral arteries | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by trans cranial Doppler
End diastolic velocity of middle cerebral arteries | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by trans cranial Doppler
Heart rate | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
Systolic blood pressure | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
Diastolic blood pressure | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
PH | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by arterial blood gases
PCo2 | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by arterial blood gases
Po2 | baseline 5 minutes after induction anesthesia,dissection phase 30 minutes after induction of anesthesia, 1 hour after drug infusion, 15 minutes after start of anhepatic phase, 5 minutes after reperfusion
  assessed by arterial blood gases

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mohamed mokhtar, M.D, Study Director — kasralainy faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czosnyka M, Brady K, Reinhard M, Smielewski P, Steiner LA. Monitoring of cerebrovascular autoregulation: facts, myths, and missing links. Neurocrit Care. 2009;10(3):373-86. doi: 10.1007/s12028-008-9175-7. Epub 2009 Jan 6. PMID 19127448
- [Background] Joshi B, Brady K, Lee J, Easley B, Panigrahi R, Smielewski P, Czosnyka M, Hogue CW Jr. Impaired autoregulation of cerebral blood flow during rewarming from hypothermic cardiopulmonary bypass and its potential association with stroke. Anesth Analg. 2010 Feb 1;110(2):321-8. doi: 10.1213/ANE.0b013e3181c6fd12. Epub 2009 Dec 11. PMID 20008083
- [Background] Dhiman RK, Kurmi R, Thumburu KK, Venkataramarao SH, Agarwal R, Duseja A, Chawla Y. Diagnosis and prognostic significance of minimal hepatic encephalopathy in patients with cirrhosis of liver. Dig Dis Sci. 2010 Aug;55(8):2381-90. doi: 10.1007/s10620-010-1249-7. Epub 2010 May 28. PMID 20508990
- [Background] Joshi B, Ono M, Brown C, Brady K, Easley RB, Yenokyan G, Gottesman RF, Hogue CW. Predicting the limits of cerebral autoregulation during cardiopulmonary bypass. Anesth Analg. 2012 Mar;114(3):503-10. doi: 10.1213/ANE.0b013e31823d292a. Epub 2011 Nov 21. PMID 22104067
- [Background] Bechstein WO, Neuhaus P. [Bleeding problems in liver surgery and liver transplantation]. Chirurg. 2000 Apr;71(4):363-8. doi: 10.1007/s001040051066. German. PMID 10840602